CLINICAL TRIAL: NCT02000908
Title: Prospective, Randomized, Double Blind Study of Photobiomodulation Therapy Using the Realief Therapy System for the Treatment of Chemotherapy-associated Peripheral Neuropathy
Brief Title: Photobiomodulation Therapy Using the Realief Therapy System for the Treatment of Chemotherapy-associated Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013LS085; WCC# 63 (Other: University of Minnesota Women's Cancer Center)
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: gynecological cancer; ovarian cancer; primary peritoneal cancer; cervical caner; peripheral neuropathy
MeSH Terms: conditions — Ovarian Neoplasms; Peripheral Nervous System Diseases | interventions — Low-Level Light Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Realief Therapy (Experimental): Each patient will be given 15-18 treatments depending on response of 30-minute duration of photobiomodulation with the Realief Therapy system, scheduled every three times weekly for 5-6 weeks. The treatments will include laser exposure of any or all of 27 differentiated areas of the legs, feet, cervical spine region and lumbar spine region, for durations of 3 to 30 minutes, based on the symptom presentation at the time. Power densities will vary from 5 to 12 watts, based on the symptom presentations through the course of therapy.
  Interventions: Device: photobiomodulation
- Sham Treatment (Sham Comparator): The placebo group will receive sham treatment, during which a heat probe will be guided over both lower extremities over a period of 30 minutes, consistent with the treatment arm. The laser device will be activated during the treatment so that the visual and auditory environment prior to therapy will be the same for both treatment and sham control.
  After 8 weeks of sham treatment the subjects in this arm will be offered the photobiomodulation combined with physiotherapy.
  Interventions: Device: photobiomodulation; Other: Sham treatment; Other: Physiotherapy

INTERVENTIONS:
Device: photobiomodulation — The photobiomodulation delivered by Realief Therapy involves amplitude wavelength light delivered by a class IV therapeutic laser.
Other: Sham treatment — All patients in sham treatment arm cross over to laser therapy followed by physiotherapy
  Arms: Sham Treatment
Other: Physiotherapy — Chiropractic massage and lymphedema treatment
  Arms: Sham Treatment

SUMMARY:
This is a 2-armed, randomized, sham-controlled, double-blinded clinical trial of photobiomodulation therapy using the Realief Therapy system. The patients will be randomized in a 3:4 ratio to treatment or sham arms.

DETAILED DESCRIPTION:
The treatments will be administered by a Realief Neuropathy Center therapist. The target surface area and treatment durations will be dictated by the Realief Therapy protocol according to their proprietary algorithm, which includes assessment of geographic areas involved and the degree of neuropathy experienced. For the trial, each patient will be given 18 treatments of 30-minute duration, scheduled every three times weekly. The treatments will include laser exposure of any or all of 27 differentiated areas of the legs, feet, cervical spine region and lumbar spine region, for durations of 3 to 30 minutes, based on the symptom presentation at the time. Power densities will vary from 5 to 12 watts, based on the symptom presentations through the course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have stable or worsening neuropathy (≥grade 2 CTCAE) after the completion of chemotherapy, with a presumptive remission. Patients who are interested in enrollment will have a baseline neuropathy assessment followed by a second evaluation 1 month later to confirm that the neuropathy is not spontaneously improving (greater than 10% improvement in their mTNS).
* Patients will be 18 years or older at the time of signing the consent.
* Patients must have GOG performance status of 0, 1, 2, or 3 (see appendix III), and be able to communicate both their symptoms and report the response to neurologic testing.
* Patients must have recovered from the acute and remediable effects of surgery, radiation therapy and/or chemoradiotherapy. At least 3 weeks must have elapsed from the last administration of chemotherapy, and at least three weeks must have elapsed from the last administration of a complete radiation therapy regimen alone or chemoradiation therapy.
* Patients with pre-existing neuropathy will be eligible, provided that they have not previously undergone laser therapy for the treatment of their condition.
* Patients must be sterile or on adequate birth control.
* Patients must have willingly signed an approved consent form, be willing to be randomized to intervention or sham therapy, and be willing to be blinded from directly observing therapy. Patients completing sham therapy will be offered Realief Therapy in conjunction with physiotherapy free of charge.
* Patients must be able to attend therapy at the Realief Neuropathy Center in St. Louis Park as dictated by the requirements of the protocol (3 times/week for up to 8 weeks as well as once 8 weeks following the completion of therapy) AND be evaluated at the University of Minnesota's Gynecologic Cancer Clinic for study assessments (4 planned assessments during and after therapy). Every effort will be made to co-ordinate these visits with routine health maintenance.
* Life expectancy >6 months

Exclusion Criteria:

* Patients who have previously received a laser-based therapy for the treatment of neuropathy will be considered ineligible.
* Patients with a > 10% improvement from the initial mTNS assessment to the mTNS assessment at the time of study enrollment (four weeks from the original assessment).
* Patients with evidence of direct tumor involvement of the nervous system (central or peripheral) will be considered ineligible.
* Patients who are pregnant will be considered ineligible. Class 4 lasers have been inadequately studied in this setting to conclude that there is no risk to a developing fetus.
* Patients with the inability to tolerate therapy or blinding due to co-morbid medical or psychiatric illness.
* Patients in active treatment of cancer will not be considered eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01-07 (Actual); Study Completion 2017-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Argenta, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Gynecologic Cancer Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Treatment: The placebo group will receive sham treatment, during which a heat probe will be guided over both lower extremities over a period of 30 minutes, consistent with the treatment arm. The laser device will be activated during the treatment so that the visual and auditory environment prior to therapy will be the same for both treatment and sham control.
  After 8 weeks of sham treatment the subjects in this arm will be offered the photobiomodulation combined with physiotherapy.
  photobiomodulation: The photobiomodulation delivered by Realief Therapy involves amplitude wavelength light delivered by a class IV therapeutic laser.
  Sham treatment: All patients in sham treatment arm cross over to laser therapy followed by physiotherapy
  Physiotherapy: Chiropractic massage and lymphedema treatment
Period: Overall Study
Arm/Group | Realief Therapy | Sham Treatment
Started | 30 | 40
Completed | 28 | 36
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Realief Therapy | Sham Treatment | Total
Number analyzed (Participants) | 30 | 40 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 30 | 39
  >=65 years | 21 | 10 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 40 | 70
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 29 | 38 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 40 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change of Total Neuropathy Score
Description: For each patient, we will compute the difference between the total neuropathy score at 8 weeks (the end of treatment) and the total neuropathy score at the time of randomization. The mean change in score for the experimental group patients will be compared to the mean change in score for the control group patients using a two-sample t-test.
  Scale scoring is 0-<20 0 being no pain <20 =severe
Time Frame: Baseline 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Realief Therapy | Sham Treatment
Number analyzed (Participants) | 30 | 38
units on a scale | -6.8 (52.6) | 0.2 (1.5)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Realief Therapy | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/40
Other Adverse Events (participants affected / at risk) | 0/30 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Realief Therapy (N=30) | Sham Treatment (N=40)
Superficial Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No